CLINICAL TRIAL: NCT02775513
Title: Metabolism of Patients With Genetically Caused Cardiac Arrhythmia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Signe Torekov, Associate professor, University of Copenhagen
Other Study IDs: LQTS
Record Dates: First submitted 2016-03-16; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mutation: Patients with functional mutation in ion channels
- Control: Matched control

SUMMARY:
Loss-of-function mutations in voltage-gated potassium channels cause long QT syndrome (LQTS) due to a prolonged cardiac repolarisation phase. Hypoteses: patients with loss-of-function mutations also exhibit altered hormone release upon glucose ingestion.

DETAILED DESCRIPTION:
Loss-of-function mutations in voltage-gated potassium channels cause long QT syndrome (LQTS) due to a prolonged cardiac repolarisation phase.

Voltage-gated potassium (Kv-) channels are known for their relation to malignant cardiac arrhythmias, but also play a role in pancreatic alpha- and beta cell hormone secretion, and possibly in incretin hormone secretion. We hypothesised that patients with loss-of-function mutations also exhibit altered hormone release upon glucose ingestion.

ELIGIBILITY:
Inclusion Criteria:

LQTS Gain of function Matched healthy controls

Exclusion criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with functional mutations in ion channels and matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
glucose homeostasis | 6 hours
  measured by glucose, insulin, glucagon, GLP-1 and GIP response to glucose (OGTT)

SECONDARY OUTCOMES:
QT | 6 hours
  cardiac repolarisation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hylten-Cavallius L, Iepsen EW, Wewer Albrechtsen NJ, Svendstrup M, Lubberding AF, Hartmann B, Jespersen T, Linneberg A, Christiansen M, Vestergaard H, Pedersen O, Holst JJ, Kanters JK, Hansen T, Torekov SS. Patients With Long-QT Syndrome Caused by Impaired hERG-Encoded Kv11.1 Potassium Channel Have Exaggerated Endocrine Pancreatic and Incretin Function Associated With Reactive Hypoglycemia. Circulation. 2017 May 2;135(18):1705-1719. doi: 10.1161/CIRCULATIONAHA.116.024279. Epub 2017 Feb 24. PMID 28235848